CLINICAL TRIAL: NCT02891616
Title: Early Assessment of Response to Dual Checkpoint Inhibitor Therapy in Patients With Advanced Melanoma Using 18F-FLT PET/CT and PET/MR
Brief Title: 18F-FLT PET Imaging in Patients With Advanced Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 201602062
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Melanoma
Keywords: Melanoma; 18F-FLT; 18F-FDG; PET/CT; PET/MR
MeSH Terms: conditions — Melanoma | interventions — Fluorodeoxyglucose F18; Positron Emission Tomography Computed Tomography; alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- FDG-PET/CT + FLT-PET/CT + PET/MR (Experimental): -Baseline, Week 3 (between days 14-20), Week 6 (between days 35-41)
  * FDG-PET/CT - Patients required to fast for at least 4 hours prior to FDG administration. Roughly 60 minutes prior to PET/CT imaging, FDG will be administered via IV bolus injection. A CT will be performed immediately before PET imaging. Whole body PET imaging will be performed for a total of about 30 minutes.
  * FLT-PET/CT - Patients required to fast for at least 4 hours prior to FLT administration. Roughly 80 minutes prior to PET/CT imaging, FLT will be administered via IV bolus injection. A CT will be performed immediately before PET imaging. Whole body PET imaging will be performed for a total of about 30 minutes.
  * PET/MR - A limited whole body scan performed immediately following PET/CT imaging when possible. Should be performed at least once at each time-point. This scan will be of a more limited area and be performed for no more than 30 minutes.
  Interventions: Drug: fludeoxyglucose F 18; Device: Positron emission tomography-computed tomography; Drug: 18F-fluorothymidine; Device: Positron emission tomography-magnetic resonance imaging

INTERVENTIONS:
Drug: fludeoxyglucose F 18
  Other Names: Fludeoxyglucose (18F); FDG
Device: Positron emission tomography-computed tomography
  Other Names: PET/CT
Drug: 18F-fluorothymidine
  Other Names: FLT
Device: Positron emission tomography-magnetic resonance imaging
  Other Names: PET/MRI; PET/MR

SUMMARY:
In the current study, advanced positron emission tomography/computed tomography (PET/CT) and positron emission tomography/magnetic resonance (PET/MR) imaging methods will be used to validate our hypothesis that melanoma patients receiving Dual-Immune Checkpoint Blockade (DICB) therapy, who ultimately achieve clinical benefit, will have an increase, or "FLARE", in tumor FLT and/or FDG uptake from baseline, as seen after cycle#1 of treatment, and that after 2 cycles of treatment responders will have a decline in FLT and FDG uptake, in comparison to the patients classified as "non-responders". In addition, alterations in tumor apparent diffusion coefficient (ADC) on diffusion-weighted magnetic resonance imaging (DW/MRI) will be evaluated, expecting after cycle#1: transient reductions in ADC due to lymphocyte proliferation, increased cellularity and restriction of water movement in responding patients, with these patients tumors having increased ADC at 2 cycles into therapy associated with tumor necrosis. This study will evaluate rather early PET imaging with FLT and FDG is a useful imaging biomarker of response to DICB.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of unresectable, stage III or metastatic melanoma.
* Patients who are eligible to receive combined dual immune-checkpoint blockade therapy with ipilimumab and nivolumab, per referring oncologist.
* Life expectancy ≥ 6 months.
* Disease that is measurable. This is defined as lesions measuring at least 10mm on radiologic imaging.
* The Eastern Cooperative Oncology Group (ECOG) performance status of 1 or better
* Age ≥18 years.
* Normal organ and marrow function as defined below

  * Aspartate aminotransferase (AST) (SGOT) or alanine aminotransferase (ALT) (SGPT) ≤2.5 × institutional upper limit of normal (≤5 x upper limit of normal for patient with liver metastasis)
  * Total bilirubin within 1.5 x institutional level of normal or direct bilirubin ≤ upper limit of normal (ULN) for patient with total bilirubin levels > 1.5 ULN)
  * Hemoglobin ≥ 9.0g/dL or ≥5.6mmol/L
  * Absolute neutrophil count ≥1000/mcL
  * Platelets ≥ 75K/mcL
* Women of child-bearing potential must have a negative urinary or serum pregnancy test within 7 days of baseline imaging.

Exclusion Criteria:

* Patient may not be receiving any other investigational agents
* Significant auto-immune disease requiring hospitalization within the past two years or any history of life-threatening auto-immune disease
* Immunosuppressive therapy including systemic corticosteroids except for maintenance dosing for adrenal insufficiency
* Known additional malignancy that is progressing or requires active treatment with the exceptions of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Active autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents with the exceptions of replacement dose steroids for adrenal insufficiency, vitiligo, resolved childhood asthma/atopy, intermittent use of inhaled steroids, local steroid injections, hypothyroidism stable on hormone replacement, and Sjogren's syndrome
* Active tuberculosis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, autoimmune diseases, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with a pacemaker, stainless steel aneurysm clip or any other magnetic resonance (MR) contraindicated implant or foreign body would warrant exclusion from this study. Pacemakers may be reprogrammed or turned off by the strong MRI magnetic field. Radio-frequency (RF) fields in MR can also cause severe heating of pacemaker lead tips. Steel aneurysm clips are prone to torque in the strong MR field which can displace the clips and may damage the vessel, resulting in hemorrhage, and/or death.
* History of pneumonitis requiring hospitalization or systemic immune suppressive therapy.
* Pregnant women are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Mean difference in FLT uptake between responders and non-responders | Baseline and Week 3
Mean difference in FLT uptake between responders and non-responders | Baseline and Week 6

SECONDARY OUTCOMES:
Mean difference in FDG uptake between responders and non-responders | Baseline and Week 3
Mean difference in FDG uptake between responders and non-responders | Baseline and Week 6
Change in ADC on DW-MRI | Baseline and Week 3
Change in ADC on DW-MRI | Baseline and Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Wahl, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu